CLINICAL TRIAL: NCT02989974
Title: Kentucky LEADS Lung Cancer Survivorship Care Program - Survivors and Caregivers
Brief Title: Kentucky LEADS Collaborative: Lung Cancer Survivorship Care Program
Acronym: KYLEADS-SC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jamie Studts (Other)
Collaborators: University of Louisville (Other); Lung Cancer Alliance (Unknown); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Jamie Studts, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-BS-01; 16-0813 (Other: Univ of KY IRB)
Record Dates: First submitted 2016-12-02; First posted 2016-12-12 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Lung Cancer
Keywords: Survivorship Care; Caregiving
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KY LEADS Survivorship Care - Survivor (Experimental): The KY LEADS Survivorship Care condition involves providing a targeted and tailored psychosocial support intervention to individuals diagnosed with lung cancer (survivor).
  Interventions: Behavioral: KY LEADS Survivorship Care
- KY LEADS Survivorship Care - Caregiver (Experimental): The KY LEADS Survivorship Care condition involves providing a targeted and tailored psychosocial support intervention to caregivers of individuals diagnosed with lung cancer (caregiver)
  Interventions: Behavioral: KY LEADS Survivorship Care

INTERVENTIONS:
Behavioral: KY LEADS Survivorship Care — Survivor: Survivor questionnaire 1 at enrollment; KY LEADS Survivorship Care Program; survivor questionnaire 2 one week after program completion; survivor questionnaire 3 six months after enrollment.
  Caregiver: Caregiver questionnaire 1 at enrollment;KY LEADS Survivorship Care Program; caregiver questionnaire 2 one week after program completion; caregiver questionnaire 3 six months after enrollment

SUMMARY:
The objective of the Kentucky LEADS Lung Cancer Survivorship Care Program is to develop, administer and evaluate the impact of a comprehensive psychosocial survivorship care program for individuals diagnosed with lung cancer and their caregivers to improve lung cancer survivorship and delivery of high-quality lung cancer care. The investigators hypothesize that the Kentucky LEADS Lung Cancer Survivorship Care Program will demonstrate improved quality of life, better symptom control, increased tobacco treatment, and reduced distress among lung cancer survivors and their caregivers.

DETAILED DESCRIPTION:
The study design is a single-arm clinical trial, or a prospective cohort design, where a longitudinal series of data will be collected from participants. Participants will be consented and asked to complete a baseline questionnaire (PRE) which includes topics measuring quality of life, distress, symptom management, social support, healthy behaviors, demographics and health history. Two similar questionnaires will be administered after exposure to the Survivorship Care Program (POST and FOL). In addition, the consent form requests permission from survivors to collect clinical data from medical records and the Kentucky Cancer Registry regarding diagnosis and treatment for lung cancer. The study will enroll 300 participants, with an estimate of approximately 30 participants enrolled at each site. However, if a participating site enrolls 30 participants and the overall study accrual has not yet been met, the study PI may allow that respective participating site to continue to enroll participants. Study accrual is competitive across participating sites until the overall study accrual has been met.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have been diagnosed with lung cancer (survivor) or
* Caregiver of a participating lung cancer survivor
* Ability to read and write in English

Exclusion Criteria:

* Individuals with significant psychiatric disturbance that requires a higher level of care
* Individuals with substance abuse/dependence problem that require a higher level of care
* Incarcerate individuals or individuals detained within the legal system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Primary Survivor Acceptability A: Percentage of participating survivors that would recommend the program to other survivors on POST survey | 1 week post-intervention up to 1 month post-intervention
  Participating survivor intervention acceptability (1A)
Primary Survivor Acceptability B: Mean rating of participating survivor intervention satisfaction on POST survey | 1 week post-intervention up to 1 month post-intervention
  Participating survivor intervention satisfaction (1B)
Primary Survivor Acceptability C: Percentage of planned intervention modules completed by participating survivors based on SC Specialists intervention delivery tracking data | 1 week post-intervention up to 1 month post-intervention
  Participating survivor intervention uptake (1C)

SECONDARY OUTCOMES:
Secondary Intervention Feasibility A: Intervention accrual rate | 6 months post-baseline
  Intervention Feasibility - study accrual rate (2A)
Secondary Intervention Feasibility B: Survivorship Care (SC) Specialist ratings of intervention feasibility based on SC Specialist ratings on POST survey | 6 months post-baseline
  Intervention Feasibility - SC Specialist ratings (2B)

OTHER OUTCOMES:
Tertiary Study Feasibility A: Questionnaire 2 survey completion rate by survivors | 1 week post-intervention up to 1 month post-intervention
  Study Feasibility - Survivor survey completion rate (3A)
Tertiary Study Feasibility B: Study drop-out rate among participating survivors | 1 week post-intervention up to 1 month post-intervention
  Study Feasibility - Survivor drop-out rate (3B)
Tertiary Study Feasibility C: Rate of missing survivor/caregiver data | 1 week post-intervention up to 1 month post-intervention
  Study Feasibility - Rate of missing survivor/caregiver data (3C)
Additional Study Efficacy A1: Survivor quality of life | 1 week post-intervention up to 1 month post-intervention
  Study Efficacy - Impact on survivor quality of life (FACT-G) (4A1)
Additional Study Efficacy B1: Survivor lung cancer specific quality of life | 1 week post-intervention up to 1 month post-intervention
  Study Efficacy - Impact on survivor lung cancer specific quality of life (FACT-L) (4B1)
Additional Study Efficacy A2: Caregiver quality of life | 1 week post-intervention up to 1 month post-intervention
  tudy Efficacy - Impact on caregiver quality of life (C-QoL) (4A2)
Additional Study Efficacy B2: Caregiver self-efficacy | 1 week post-intervention up to 1 month post-intervention
  Study Efficacy - Impact on caregiver self-efficacy (CSES) (4B2)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie L Studts, PhD, Principal Investigator — Professor, University of Kentucky College of Medicine
Locations (9):
- United States (9):
  - Kings Daughters Medical Center - Ashland, Ashland, Kentucky
  - Commonwealth Cancer Center - Danville, Danville, Kentucky
  - Hardin Memorial Health - Elizabethtown, Elizabethtown, Kentucky
  - Hazard ARH Regional Medical Center, Hazard, Kentucky
  - Markey Cancer Center, Lexington, Kentucky
  - UofL/Brown Cancer Center - Louisville, Louisville, Kentucky
  - Baptist Health - Madisonville, Madisonville, Kentucky
  - St. Claire Regional Medical Center - Morehead, Morehead, Kentucky
  - Owensboro Health, Owensboro, Kentucky

IPD SHARING:
Plan to Share IPD: No